CLINICAL TRIAL: NCT02441582
Title: The Effect of 12 Lead ECG Telemetry on Reperfusion Time in Resource-limited Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: ER24 (Unknown); University of Stellenbosch (Other); Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Willem Stassen, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 3-1178/2014
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Infarction; STEMI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Telemetry

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemetry (Experimental): In this group, participants will have a prehospital 12 lead ECG taken and sent through to the receiving facility.
  Interventions: Other: Telemetry
- Non-Telemetry (Other): In this group, participants will have a prehospital 12 lead ECG taken which will not be sent through to the receiving facility.
  Interventions: Other: Non-telemetry

INTERVENTIONS:
Other: Telemetry
  Arms: Telemetry
Other: Non-telemetry
  Arms: Non-Telemetry

SUMMARY:
This study aims to determine whether prehospital 12 lead ECG telemetry decreases the time to reperfusion in patients presenting with STEMI. A randomised controlled trial will be conducted in Gauteng and the Western Cape among 100 adult patients (>18 years) presenting with ST-elevation myocardial infarction according to a specific inclusion and exclusion criteria outlined in the full protocol. Consenting patients will be randomly assigned to have their prehospital ECG sent to the receiving cardiac facility or not. The onset-to-reperfusion and door-to-reperfusion times will be recorded and compared between the two groups by using the Fisher's exact test and a simple unpaired Student's t-test. Data will also be subjected to multivariate analysis of variance to test for statistical significance within a variety of factors that may influence reperfusion times.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years of age)
* Patients presenting within the Gauteng or Western Cape areas
* Current chest pain or dyspnoea, presumed to be of cardiac origin
* ST-elevation (STEMI) on the ECG (defined as ST-elevation of 0.1 mV in two or more contiguous leads).

Exclusion Criteria:

* Non-adult patients
* Chest pain of non-cardiac aetiology (following trauma or due to a primary respiratory pathology)
* Non-consent to inclusion within the study
* Patients without medical aid or who states that they cannot afford private healthcare.
* Non-ST-elevation myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Reperfusion Time | At the first moment of reperfusion, from the date of randomisation up to 14 days
  This outcome measures the time it takes to reperfuse a coronary artery in STEMI

SECONDARY OUTCOMES:
Prehospital Time | On arrival at hospital; from the time of randomisation up to six hours
  The prehospital time is the total time from arrival at the patient to arrival at the hospital
Onset to reperfusion time | At the first moment of reperfusion, from the date of randomisation up to 14 days
  This pertains to the time it takes from the moment of first onset of symptoms to the first moment of reperfusion

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - ER24 Gauteng Region, Johannesburg, Gauteng
  - ER24 Western Cape Region, Cape Town, Western Cape